CLINICAL TRIAL: NCT00027859
Title: A Phase III Randomized Trial for Evaluating Second Line Hormonal Therapy (Ketoconazole/Hydrocortisone) Versus Paclitaxel/Estramustine Combination Chemotherapy on Progression Free Survival in Asymptomatic Patients With a Rising PSA After Hormonal Therapy for Prostate Cancer
Brief Title: Hormone Therapy Compared With Combination Chemotherapy in Treating Patients With Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); SWOG Cancer Research Network (Network); Cancer and Leukemia Group B (Network)
Responsible Party: Group Chair, Eastern Cooperative Oncology Group
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000069088; E1899; SWOG-E1899; CALGB-E1899
Record Dates: First submitted 2001-12-07; First posted 2003-01-27 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage III prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Estramustine; Ketoconazole; Hydrocortisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: docetaxel
Drug: estramustine phosphate sodium
Drug: ketoconazole
Drug: therapeutic hydrocortisone

SUMMARY:
RATIONALE: Androgens can stimulate the growth of prostate cancer cells. Drugs such as ketoconazole may stop the production of androgens. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known whether hormone therapy is more effective than combination chemotherapy in treating prostate cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of hormone therapy with that of combination chemotherapy in treating patients who have prostate cancer that has been previously treated with androgen suppression.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare time to objective progression in patients with prostate cancer and a rising prostate-specific antigen (PSA) after androgen suppression when treated with second-line hormonal therapy (ketoconazole and hydrocortisone) vs combination chemotherapy (docetaxel and estramustine).
* Compare time to PSA progression and correlate this with time to objective progression in patients treated with these regimens.
* Compare the quality of life in patients treated with these regimens.
* Compare overall survival of patients treated with these regimens.
* Compare the natural history of progression in patients treated with these regimens.
* Identify prognostic indicators of clinical outcome by immunohistochemical evaluation of apoptopic biomarkers in patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to prior treatment with bisphosphonates (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral ketoconazole three times daily and oral hydrocortisone twice daily. Treatment continues in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive oral estramustine three times daily on days 1-5 and docetaxel IV over 1 hour on day 2. Treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, on day 1 of week 9, at 6 months and 1 year, and then annually for up to 10 years or until beginning of first non-protocol therapy.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually for 5 years.

PROJECTED ACCRUAL: A total of 590 patients (295 per treatment arm) will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate that was continuously treated with androgen suppression
* Rising prostate-specific antigen (PSA), defined as PSA > 5 ng/mL, rising on 2 consecutive measurements at least 4 weeks apart
* Gleason score 7 or higher and/or seminal vesicle involvement at diagnosis
* Patients previously treated with antiandrogen or glucocorticoid therapy must meet the following criteria:

  * Must show a continued rise in PSA after stopping antiandrogen (flutamide, bicalutamide, or nilutamide) or glucocorticoid (dexamethasone or prednisone)

    * At least 4 weeks continued rise in PSA after flutamide or nilutamide (6 weeks for bicalutamide)
* Testosterone less than 50 ng/dL

  * Patients who have not undergone surgical castration must continue primary androgen suppression to maintain castrate levels of testosterone
* No progressive or measurable local or metastatic disease (including bone metastases)

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Granulocyte count at least 2,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* SGOT no greater than 2 times upper limit of normal
* Bilirubin no greater than 1.5 mg/dL

Renal:

* Creatinine no greater than 1.7 mg/dL

Cardiovascular:

* No American Heart Association class III or IV heart disease
* No uncontrolled congestive heart failure
* No life-threatening cardiac arrhythmias

Other:

* Fertile patients must use effective contraception
* No other prior malignancy unless curatively treated and disease-free for appropriate time period for specific cancer
* No preexisting peripheral neuropathy greater than grade 1
* No known hypersensitivity to polysorbate 80

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 5 years since prior systemic chemotherapy

Endocrine therapy:

* See Disease Characteristics
* At least 4 weeks since prior hydrocortisone
* No prior ketoconazole

Radiotherapy:

* At least 28 days since prior radiotherapy to primary site
* No prior palliative radiotherapy
* No concurrent radiotherapy

Surgery:

* See Disease Characteristics

Other:

* Recovered form prior therapy
* At least 7 days since prior parenteral antibiotics for active infection
* No concurrent digitalis
* No concurrent H_2 blockers or proton pump inhibitors (arm I only)
* Concurrent bisphosphonates allowed provided they were initiated prior to study therapy

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-10-08 (Actual); Primary Completion 2004-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael A. Carducci, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins; Nirmala Bhoopalam, MD, Study Chair — Veterans Affairs Medical Center - Hines; Gregory P. Swanson, MD, Study Chair — Deaconess Medical Center, Spokane, Washington; William Dahut, MD, Study Chair — National Cancer Institute (NCI)
Locations (98):
- United States (98):
  - Comprehensive Cancer Institute, Huntsville, Alabama
  - CCOP - Mayo Clinic Scottsdale Oncology Program, Scottsdale, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Veterans Affairs Medical Center - Little Rock, Little Rock, Arkansas
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Cedars-Sinai Comprehensive Cancer Center at Cedars-Sinai Medical Center, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - Naval Medical Center - San Diego, San Diego, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Medical Center of Aurora - South Campus, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - Rocky Mountain Cancer Centers - Denver Rose, Denver, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Incorporated, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - St. Mary-Corwin Regional Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Thornton, Thornton, Colorado
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Memorial Regional Cancer Center at Memorial Regional Hospital, Hollywood, Florida
  - H. Lee Moffitt Cancer Center and Research Institute at University of South Florida, Tampa, Florida
  - Veterans Affairs Medical Center - Tampa (Haley), Tampa, Florida
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Veterans Affairs Medical Center - Hines, Hines, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - West Suburban Center for Cancer Care, River Forest, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Veterans Affairs Medical Center - Indianapolis (Roudebush), Indianapolis, Indiana
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Veterans Affairs Medical Center - New Orleans, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Lakeland Cancer Care Center at Lakeland Hospital - St. Joseph, Saint Joseph, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - New Hampshire Oncology-Hematology, PA - Hooksett, Hooksett, New Hampshire
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - Cape Fear Valley Health System, Fayetteville, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Goldsboro, North Carolina
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Abramson Cancer Center at the University of Pennsylvania, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Veterans Affairs Medical Center - Charleston, Charleston, South Carolina
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - Vanderbilt-Ingram Cancer Center at Vanderbilt Medical Center, Nashville, Tennessee
  - Harrington Cancer Center, Amarillo, Texas
  - Veterans Affairs Medical Center - Amarillo, Amarillo, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - Martha Jefferson Hospital, Charlottesville, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Incorporated - Roanoke, Roanoke, Virginia
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - St. Mary's Medical Center, Huntington, West Virginia
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin

REFERENCES:
- [Result] Walczak JR, Carducci MA; Eastern Cooperative Oncology Group E1899. Phase 3 randomized trial evaluating second-line hormonal therapy versus docetaxel-estramustine combination chemotherapy on progression-free survival in asymptomatic patients with a rising prostate-specific antigen level after hormonal therapy for prostate cancer: an Eastern Cooperative Oncology Group (E1899), Intergroup/Clinical Trials Support Unit study. Urology. 2003 Dec 29;62 Suppl 1:141-6. doi: 10.1016/j.urology.2003.09.006. PMID 14747052